CLINICAL TRIAL: NCT06511349
Title: Clinical Exploration Study of YOLT-203 in the Treatment of Type 1 Primary Hyperoxaluria (PH1)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH1-YOLT-203-001
Record Dates: First submitted 2024-07-04; First posted 2024-07-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Primary Hyperoxaluria
MeSH Terms: conditions — Primary hyperoxaluria type 1

STUDY DESIGN:
Intervention Model Description: 0.3mg/kg,0.45mg/kg,0.6mg/kg,35mg
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOLT-203 (Experimental)
  Interventions: Drug: YOLT-203

INTERVENTIONS:
Drug: YOLT-203 — The IP is administered intravenously at the predetermined dose.

SUMMARY:
This study is a single-arm, open-label, single-dose, dose-escalation, and dose-expansion trial, aiming to assess the safety and tolerability of YOLT-203 in Chinese patients with Primary Hyperoxaluria Type 1 (PH1), and to preliminarily evaluate the effect of a single dose of YOLT-203 on plasma oxalate levels.

In this study, the maximum duration of the screening period is 60 days, with the treatment day being Day 1 (D1), and the safety follow-up period extending to the 52nd week after dosing. Additionally, in the dose-escalation phase, after the first dose cohort, investigators will conduct a comprehensive evaluation based on safety, pharmacokinetic (PK), and pharmacodynamic (PD) data, and following discussion at the Safety Review Committee (SRC) meeting, subjects may voluntarily receive a second administration of the study drug at an effective dose level.

After the completion of the main study, subjects will undergo long-term follow-up. In accordance with the requirements of the "Technical Guidance for Clinical Research on Long-term Follow-up of Gene Therapy Products (Trial)" issued by the Center for Drug Evaluation (CDE), long-term follow-up will be conducted for up to 15 years after dosing.

DETAILED DESCRIPTION:
As of December 2024, the clinical study of YOLT-203 for the treatment of type 1 primary hyperoxaluria (PH1) has completed enrollment and dosing for two cases at 0.3mg/kg and three cases at 0.45mg/kg, as well as a 28-day follow-up for all participants. On December 6, 2024, a meeting was held to discuss the safety and efficacy data of all participants in the two dosage groups and to make decisions on the next steps of the research plan.

Based on the safety and efficacy data from all participants in this project, the sponsor and investigators reached a consensus after a meeting discussion: YOLT-203 has good safety, and 0.45mg/kg is the anticipated biologically effective dose (OBD). According to the protocol design, the meeting decision was made to stop dose escalation and repeat a group at the anticipated effective dose (0.45mg/kg), continuing to enroll 1-3 more participants for exploratory studies.

ELIGIBILITY:
Inclusion Criteria:

* The age is ≥ 2 years old at the time of signing the informed consent.
* Have AGXT gene mutations and be diagnosed with primary hyperoxaluria (PH1); eGFR ≥ 30 ml/min/1.73m2.
* At least 2 times of 24-hour urinary oxalate excretion ≥ 0.7 mmol/1.73m2/day or the ratio of urinary oxalate to creatinine in a single urine collection must be higher than the upper limit of normal (ULN) for the corresponding age.
* If treated with vitamin B6, the treatment has been stable for 90 days before enrollment in the study and is willing to maintain the stable treatment plan unchanged during the study.
* The patient himself/herself or the guardian voluntarily signs the informed consent.

Exclusion Criteria:

* The investigator judges that there is clinical evidence of systemic extra-renal oxalate deposition.
* Have any of the following laboratory parameter assessment results at screening:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x the upper limit of normal (ULN).
  2. Total bilirubin > 1.5 x ULN. If the increase in total bilirubin is caused by diagnosed Gilbert's syndrome and the total bilirubin < 2 x ULN, it is eligible.
  3. International normalized ratio (INR) > 1.5 (Patients on oral anticoagulants [such as warfarin] and with INR < 3.5 will be allowed to participate).
* Known to have active human immunodeficiency virus (HIV) infection; or have evidence of current or chronic hepatitis C virus (HCV) or hepatitis B virus (HBV) infection.
* The estimated glomerular filtration rate (GFR) at screening is less than 30 mL/min/1.73m² (For patients ≥ 18 years old, it will be calculated according to the Modification of Diet in Renal Disease [MDRD] formula; for patients < 18 years old, it will be calculated according to the Schwartz bedside formula). See the attachment.
* Have received an investigational drug within the last 30 days or 5 half-lives (whichever is longer) before the first administration of the study drug, or have participated in the follow-up of another clinical study before randomization.
* Have a history of kidney or liver transplantation.
* According to the investigator's opinion, have other medical conditions or comorbidities that may interfere with study compliance or data interpretation.
* Have a history of multiple drug allergies or allergic reaction history to oligonucleotides or LNP.
* Have a history of subcutaneous injection intolerance.
* Unwilling to comply with contraceptive requirements throughout the study participation period until 6 months after the end of the main study trial.
* Female patients are pregnant, planning to become pregnant or breastfeeding.
* Unwilling or unable to limit alcohol consumption throughout the study. Alcohol consumption during the study exceeds 2 units per day (1 unit: approximately 125 ml of wine = approximately 29 ml of spirits = approximately 284 ml of beer, will be excluded.
* The investigator believes that there is a history of alcohol abuse within 12 months before screening.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | through week 52
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
pharmacokinetics of YOLT-203 | through Day 14
  The Peak Plasma Concentration (Cmax) of YOLT-203. 0.5 predose,2,6,24,48,72,144,312 hours
pharmacokinetics of YOLT-203 | through Day 14
  Area under the plasma concentration versus time curve (AUC). 0.5 predose,2,6,24,48,72,144,312 hours
pharmacokinetics of YOLT-203 | through Day 28
  Tmax
pharmacokinetics of YOLT-203 | through Day 28
  T1/2
pharmacodynamics | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in blood glycolic acid levels
pharmacodynamics | through week 52
  After medication, at 2, 8, 16, 24, and 52 weeks, the changes in 24-hour urinary oxalic acid excretion compared to the baseline value.
pharmacodynamics | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in 24-hour urinary glycolic acid excretion
pharmacodynamics | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in eGFR.

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China